CLINICAL TRIAL: NCT07122921
Title: Sleep Disturbance in Hong Kong Children With Cancer: A Cross-Sectional Study Comparing Healthy Counterparts and Children With Other Chronic Diseases
Brief Title: Cross-sectional Study of Sleep Disturbance in Hong Kong Children With Cancer Comparing With Healthy Counterparts and Children With Other Chronic Diseases
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mak Shuk Yan, Principal Investigator, Ward Manager (Paed), Chinese University of Hong Kong
Other Study IDs: PAED-2025-045
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Sleep; Sleep Disturbances in Children; Sleep Disturbances
Keywords: sleep; sleep disturbance; children; paediatrics
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control: The healthy control group will be of adequate sample size. These include siblings of pediatric patients (both oncology and non-oncology wards), and children of hospital staff (e.g., nurses, administrative personnel). Inclusion criteria require no history of chronic illness, psychiatric disorders, or known sleep conditions. Parental consent and child assent will be obtained for all participants.
- Children with Other Chronic Illnesses: This group will comprise children diagnosed with chronic conditions other than cancer, such as asthma, type 1 diabetes, or chronic kidney disease, recruited from the cardiac, nephrology, and mixed wards of Hong Kong Children's Hospital. These illnesses are selected for their known potential to disrupt sleep-e.g., nocturnal asthma symptoms or glucose instability-while differing in pathophysiology from cancer. Participants must be under active management for their condition and currently hospitalized, but must not have a history of primary sleep disorders (e.g., narcolepsy, obstructive sleep apnea) unrelated to their chronic illness. This criterion ensures that observed sleep disturbances are attributable to the chronic condition rather than pre-existing sleep pathology.
- Children with Cancer: Participants in this group will be children with a confirmed cancer diagnosis, such as leukemia, lymphoma, or solid tumors, who are currently hospitalized for treatment at the inpatient oncology wards of Hong Kong Children's Hospital. Eligible participants must be actively receiving cancer-directed therapy (e.g., chemotherapy, radiation) during their hospital stay. Inclusion criteria require that participants, or their parents or legal guardians as proxies, can provide accurate reports about sleep patterns, either through self-assessment or observation, ensuring reliable data collection. This group will capture the acute impact of cancer treatment and hospitalization on sleep, a critical focus of the study.

SUMMARY:
Sleep disturbances are prevalent among children with chronic illnesses, yet the specific impact of cancer on sleep remains underexplored. This prospective and cross-sectional study aims to evaluate the prevalence, severity, and characteristics of sleep disturbances in Chinese children with cancer compared to healthy peers and children with other chronic diseases. By leveraging validated sleep assessment tools and parental reports, the goal is to identify unique challenges faced by children with cancer. Results might influence the design of personalized interventions aimed at enhancing the overall well-being of children with cancer.

This study will enroll Chinese children aged 6 to 18 years, divided into three distinct groups based on their health status: children with cancer, children with other chronic illnesses, and healthy children. A total sample size of 150 participants (50 per group) will be targeted to ensure adequate statistical power for comparative analyses. Recruitment will occur at Hong Kong Children's Hospital or the cancer and chronic illness groups, and healthy children will be recruited from healthy siblings of participants or the healthy children of hospital staff with specific inclusion and exclusion criteria applied to each group to maintain homogeneity and minimize confounding variables.

DETAILED DESCRIPTION:
The objectives of this study are threefold:

1. To assess the prevalence and nature of sleep disturbances in children with cancer.
2. To compare sleep disturbances in children with cancer to those in healthy children and children with other chronic diseases.
3. To identify potential factors contributing to sleep disturbances in paediatric patients.

Sleep quality, measured by the global PSQI score, will be the primary endpoint. This encompasses the seven component scores (e.g., sleep duration, latency, efficiency), providing a holistic assessment of sleep health. A global score >5 will classify participants as having poor sleep quality, enabling prevalence comparisons across groups.

Health-related quality of life, assessed via the PedsQL total score and its domain-specific subscales (physical, emotional, social, school), as well as physical health summary score and psychosocial health summary score will examine the broader impact of sleep disturbances. This will help determine, for example, whether poor sleep in children with cancer correlates with reduced emotional or physical functioning compared to other groups.

To control for potential confounding effects on sleep patterns and access to healthcare resources, the following demographic and clinical variables will be collected: age (in years), gender, socioeconomic status (SES), disease type, disease status, and use of hypnotics (yes/no). SES will be assessed through parental education (categorized as primary or below, junior secondary, senior secondary, or university/college and above). For children with cancer, disease type (e.g., leukemia, lymphoma, brain tumor, bone tumor, or others) and disease status (e.g., stage 1-4, recurrence, years since diagnosis, treatment type such as chemotherapy, radiotherapy, surgery, immunotherapy, transplant, or combination) will be recorded. For children with other chronic illnesses, disease type (e.g., asthma, type 1 diabetes, chronic kidney disease) will be noted. These factors may influence sleep outcomes, e.g., older children may report greater daytime dysfunction, or lower parental education level may limit access to supportive care, necessitating adjustment in statistical analyses to isolate the effects of chronic illness on sleep quality.

This study anticipates uncovering significant differences in sleep quality between children hospitalized with cancer, those with other chronic illnesses, and healthy children. The following outcomes are expected:

1. It is hypothesized that children with cancer will exhibit the most severe sleep disturbances among the three groups. Factors such as pain associated with the illness, side effects of chemotherapy, and frequent nighttime medical interventions are likely to result in reduced sleep duration, prolonged sleep latency, and increased sleep fragmentation. Reported data from the PSQI are also expected to place a majority of children with cancer above the clinical threshold for poor sleep.
2. While children with other chronic illnesses are also expected to experience sleep disturbances, these disruptions are likely to be less severe than those observed in children with cancer. For example, conditions such as asthma or diabetes may cause episodic sleep interruptions (e.g., nocturnal coughing or nighttime glucose monitoring), but they are not typically compounded by the environmental and psychological stressors associated with hospitalization. A smaller percentage of this group is anticipated to exceed the clinical threshold for poor sleep on the PSQI.
3. Healthy children are expected to demonstrate the highest sleep quality among the three groups, with results showing near-optimal sleep duration and efficiency. Reported data are anticipated to reflect low levels of sleep disturbances, with the majority of children scoring below the clinical threshold on the PSQI. These findings will provide a baseline for understanding how chronic illnesses and hospitalization affect sleep outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Cancer (n=50) Participants in this group will be children with a confirmed cancer diagnosis, such as leukemia, lymphoma, or solid tumors, who are currently hospitalized for treatment at the inpatient oncology wards of Hong Kong Children's Hospital. Eligible participants must be actively receiving cancer-directed therapy (e.g., chemotherapy, radiation) during their hospital stay. Inclusion criteria require that participants, or their parents or legal guardians as proxies, can provide accurate reports about sleep patterns, either through self-assessment or observation, ensuring reliable data collection. This group will capture the acute impact of cancer treatment and hospitalization on sleep, a critical focus of the study.
2. Children with Other Chronic Illnesses (n=50) This group will comprise children diagnosed with chronic conditions other than cancer, such as asthma, type 1 diabetes, or chronic kidney disease, recruited from the cardiac, nephrology, and mixed wards of Hong Kong Children's Hospital. These illnesses are selected for their known potential to disrupt sleep-e.g., nocturnal asthma symptoms or glucose instability-while differing in pathophysiology from cancer. Participants must be under active management for their condition and currently hospitalized, but must not have a history of primary sleep disorders (e.g., narcolepsy, obstructive sleep apnea) unrelated to their chronic illness. This criterion ensures that observed sleep disturbances are attributable to the chronic condition rather than pre-existing sleep pathology.
3. Healthy Children (n=50) The healthy control group will be of adequate sample size. These include siblings of pediatric patients (both oncology and non-oncology wards), and children of hospital staff (e.g., nurses, administrative personnel). Inclusion criteria require no history of chronic illness, psychiatric disorders, or known sleep conditions. Parental consent and child assent will be obtained for all participants.

Exclusion Criteria:

Across all three groups, children will be excluded if they are not Chinese and are in intensive care units. Children who exhibit severe cognitive impairments that preclude accurate reporting of sleep experiences, either by themselves or their parents or legal guardians, will be excluded. Additionally, participants with neurological conditions known to independently affect sleep, such as epilepsy or cerebral palsy, will be excluded to avoid confounding the primary relationship between chronic illness and sleep disturbances. The use of sedative medications unrelated to the participant's primary condition (e.g., for behavioral management rather than cancer treatment) will also disqualify participants, as these could artificially alter sleep patterns and obscure study outcomes. These exclusion criteria ensure that sleep disturbances observed are primarily linked to the participants' health status rather than extraneous factors.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Paediatrics
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 1 month
  Sleep quality, measured by the global PSQI score, will be the primary endpoint. This encompasses the seven component scores (e.g., sleep duration, latency, efficiency), providing a holistic assessment of sleep health. A global score >5 will classify participants as having poor sleep quality, enabling prevalence comparisons across groups.
Health-related quality of life | 1 month
  Health-related quality of life, assessed via the PedsQL total score and its domain-specific subscales (physical, emotional, social, school), as well as physical health summary score and psychosocial health summary score will examine the broader impact of sleep disturbances. This will help determine, for example, whether poor sleep in children with cancer correlates with reduced emotional or physical functioning compared to other groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No intervention involved

DOCUMENTS (1):
  • Study Protocol (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT07122921/Prot_000.pdf